CLINICAL TRIAL: NCT00548470
Title: Evaluation of Varenicline's Clinical Efficacy for Continued Smoking Abstinence When Used in the Clinical Treatment of Schizophrenic Patients Hospitalized in an Institution With a Ban on Cigarette Smoking
Brief Title: Varenicline Effects In Schizophrenic Smokers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nathan Kline Institute for Psychiatric Research (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Robert C. Smith MD PhD, Research Psychiatrist, Prinicipal Investigator, Nathan Kline Institute for Psychiatric Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06I/C34-0
Record Dates: First submitted 2007-10-22; First posted 2007-10-24 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2017-10

CONDITIONS: Schizophrenia; Tobacco Use Disorder; Nicotine Dependance
Keywords: schizophrenia; varenicline; cognition; cigarette smoking
MeSH Terms: conditions — Schizophrenia; Tobacco Use Disorder; Cigarette Smoking | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- varenicline (Experimental): open label varenicline 2mg/day
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — Varenicline 1-2 mg/day
  Other Names: Chantix

SUMMARY:
This is an open label pre-post study of the effects of clinical treatment with varenicline on 1) decreasing smoking in schizophrenic patients, 2) improving selected cognitive measures in schizophrenic patients, and 3) psychopathology in schizophrenic patients. Patients are assessed on subjective and objective measures of smoking, selected cognitive measures, and special chemical measures, during baseline testing and during 8 weeks of treatment with varenicline (1-2 mg/day).

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Schizophrenia or Schizoaffective Psychosis
* Recent History of Cigarette smoking
* Ages 18-65

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-06; Primary Completion 2009-09 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Smith, MD, PhD, Principal Investigator — Nathan Kline Institute of Psychiatric Research; NYU School of Medicine
Locations (1):
- Manhattan Psychiatric Center, New York, New York, United States

REFERENCES:
- [Result] Smith RC, Lindenmayer JP, Davis JM, Cornwell J, Noth K, Gupta S, Sershen H, Lajtha A. Cognitive and antismoking effects of varenicline in patients with schizophrenia or schizoaffective disorder. Schizophr Res. 2009 May;110(1-3):149-55. doi: 10.1016/j.schres.2009.02.001. Epub 2009 Feb 28. PMID 19251401

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenciline: open label varenicline 2mg/day
  Varenicline: Varenicline 1-2 mg/day
Period: Overall Study
Arm/Group | Varenciline
Started | 14
Completed | 12
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Varenciline
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 1
  african american | 11
  hispanic | 2
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Self Report of Smoking
Description: Patients self-report of smoking cigarettes. Patients were interviewed weekly about the number of cigarettes smoked. Number of cigarettes smoked in the past week.
Time Frame: Baseline and during 2 months of treatment
Measure: Mean (Standard Deviation); unit: Cigarettes
Arm/Group | Varenciline
Number analyzed (Participants) | 12
Cigarettes
  Cigarettes smoked baseline | 36.45 (63.03)
  Cigarettes smoked month 1 | 17.25 (29.74)
  Cigarettes smoked month 2 | 12.52 (20.11)

2. Primary Outcome: CO (Carbon Monoxide) Breathalyzer Level
Description: Carbon Monoxide in breath ,parts per million
Time Frame: baseline and during 2 months of treatment
Measure: Mean (Standard Deviation); unit: ppm (carbon monoxide parts per million)
Arm/Group | Varenciline
Number analyzed (Participants) | 12
ppm (carbon monoxide parts per million)
  CO level baseline | 8.97 (6.21)
  CO level month 1 | 5.7 (4.00)
  CO level month 2 | 4.85 (4.41)

3. Primary Outcome: Plasma Cotinine
Description: cotinine level in plasma ng/ml.
Time Frame: baseline 1 month and 2 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Varenciline
Number analyzed (Participants) | 12
ng/ml
  baseline cotinine | 362.25 (120.93)
  1 month cotinine | 181.75 (144.08)
  2 month cotinine | 200.25 (129.75)

4. Secondary Outcome: RBANS Neuropsychological Battery
Description: The scale is Repeatable Battery for the Assessment to Neuropsychological Status (RBANS). This scale measures cognitive function in patients with schizophrenia. RBANS scores for list learning range from 0 to 40. RBANS Index scores for visual-spatial index, language index, and Total score range from 40-160. RBANS Total score is the sum of score of all the individual items ( items 1-12) on the RBANS scale. List Learning scores range from 0 to 40. Visual Spatial Construction index scores range from 0 to 30.. Higher scores on all these measures indicate better performance or better cognitive ability.
Time Frame: baseline and month 2 of treatment
Measure: Mean (Standard Deviation); unit: RBANS scores
Arm/Group | Varenciline
Number analyzed (Participants) | 12
RBANS scores
  RBANS total baseline | 59.00 (13.10)
  RBANS total 2 months | 59.17 (9.26)
  RBANS l;ist learning baseline | 15.75 (5.50)
  RBANS list learning 2 months | 19.50 (4.19)
  RBANS visuospatal index baseline | 73.58 (7.44)
  RBANS visuospatial index 2 months | 63.50 (8.07)
  RBANS language index baseline | 70.17 (13.23)
  RBANS language index 2 months | 83.50 (12.55)

5. Secondary Outcome: Change From Baseline in Psychiatric Symptoms
Description: The Positive and Negative Syndrome Scale (PANSS) was used to measure psychiatric symptoms. Item scores ranged from 1 (Absent) to 6 (Severe) for symptoms on the Positive Scale (total subscale range: 7-42), the Negative Scale (total subscale range: 7-42), and the General Psychopathology Scale (total subscale range:16-96). All three subscales were summed for the PANSS total score (total scale range: 30-180). Higher numbers indicate more psychopathology. Therefore, if scores are reduced at post-baseline ratings, this would indicate lower psychopathology.
Time Frame: Baseline and 2 months later
Measure: Mean (Standard Deviation); unit: Units on the PANSS scale
Arm/Group | Varenciline
Number analyzed (Participants) | 12
Units on the PANSS scale
  PANSS total baseline | 56.57 (12.72)
  PANSS total 2 months | 55.58 (9.41)
  PANSS Positive baseline | 12.58 (5.41)
  PANSS Positive 2 months | 12.00 (5.59)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Varenicline
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 2/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=14)
nausea (Gastrointestinal disorders) | 2 (2) — nausea reported on varenicline

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No